CLINICAL TRIAL: NCT04889391
Title: A Phase I, Open-Label, Single Dose ADME Study of 14C-ACH-0144471 in Healthy Male Subjects
Brief Title: Study of Radiolabeled Danicopan in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-005
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Danicopan; ACH-0144471; ALXN2040; Absorption; Distribution; Metabolism; Excretion; Total Radioactivity; ADME
MeSH Terms: interventions — danicopan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]-Danicopan (Experimental): Participants were administered a single oral dose of danicopan between 151 and 154 mg (nominal dose of 150 mg), providing approximately 100 μCi of [14C] radiolabel in the form of [14C]-danicopan.
  Interventions: Drug: [14C]-Danicopan

INTERVENTIONS:
Drug: [14C]-Danicopan — Liquid-filled capsules.
  Other Names: ALXN2040; ACH-014447; ACH-4471; ACH4471; 4471

SUMMARY:
This was an open-label study to evaluate the absorption, distribution, metabolism, and excretion of radioactivity in healthy male participants following a single 150-milligram (mg) oral dose of carbon-14 ([14C])-ACH-014447 ([14C])-danicopan) containing approximately 100 microcuries (µCi) of [14C].

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy was defined as having no clinical relevant abnormalities identified by a detailed medical history, physical exam, blood pressure and pulse rate measurements, 12-lead electrocardiogram, and clinical laboratory tests.
* Body mass index of ≥ 18 and ≤ 30 kilograms (kg)/meter squared and weight of ≥ 50 kg and ≤ 100 kg.
* Regular daily bowel movements (that is, production of at least 1 stool per day).
* Non-smoker or ex-smoker who had not used tobacco or nicotine products for ≥ 3 months prior to screening.

Key Exclusion Criteria:

* History or clinically relevant evidence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* History of conditions or procedures possibly affecting drug absorption or excretion. A history of appendectomy, cholecystectomy, and hernia repair was allowed if they were not associated with complications.
* Active bacterial infection or clinically significant active viral infection, a body temperature > 38°Celcius, or other evidence of infection on Day 1, or with a history of febrile illness within 7 days prior to Day 1.
* Healthy participants who had been exposed to significant radiation levels of > 5 millisieverts in the last year prior to screening.
* Clinically significant laboratory abnormalities at screening or Day -1, as well as absolute neutrophil counts, platelets, and hemoglobin outside of reference ranges.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Mean Cumulative Percentages Of Total Radioactivity Recovered In Urine And Feces Following A Single Oral Dose Of [14C]-Danicopan | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
Whole Blood And Plasma Pharmacokinetics (PK) Of Total Radioactivity After A Single Oral Dose Of [14C]-Danicopan: Area Under The Concentration-time Curve From Time 0 To The Time Of Last Quantifiable Concentration (AUC0-t) | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
Whole Blood And Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-Danicopan: Area Under The Concentration-time Curve Extrapolated to Infinity (AUC0-inf) | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
Whole Blood And Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-Danicopan: Maximum Observed Concentration (Cmax) | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
Whole Blood And Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-Danicopan: Time To Maximum Observed Concentration (Tmax) | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
Plasma PK Of Danicopan After A Single Oral Dose Of [14C]-Danicopan: AUC0-t | Up to 96 hours postdose
Plasma PK Of Danicopan After A Single Oral Dose Of [14C]-Danicopan: AUC0-inf | Up to 96 hours postdose
Plasma PK Of Danicopan After A Single Oral Dose Of [14C]-Danicopan: Cmax | Up to 96 hours postdose
Plasma PK Of Danicopan After A Single Oral Dose Of [14C]-Danicopan: Tmax | Up to 96 hours postdose
[14C]-Danicopan Metabolites In Plasma, Urine, And Feces | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period

SECONDARY OUTCOMES:
Percentage Of Total Radioactivity Detected For Each [14C]-Danicopan Metabolite in Plasma, Urine, And Feces | Up to 96 hours postdose or maximum of 216 hours postdose for extended collection period
  [14C]-Danicopan metabolic profiling in plasma, urine, and feces was performed in samples containing sufficient amounts of radioactivity. The percent of dose represented by each of the metabolites was calculated using the radioactivity concentration equivalent data combined with the metabolic profiling data. The percentage of each identified metabolite to total radioactivity in plasma was estimated based on plasma metabolic profiling data.
Incidence Of Treatment-emergent Adverse Events | Day 1 through Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand